CLINICAL TRIAL: NCT06793657
Title: Poppy Seed Use in Gastroenteric Fistula Diagnosis in Gynecologic Oncology Surgery
Brief Title: Poppy Seed Use in Gastroenteric Fistula Diagnosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Albayrak, Principal Investigator, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/2142
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Gynecologic Cancers; Fistula
MeSH Terms: conditions — Fistula | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Intervention Model Description: A single arm study that will compare computed tomography and oral poppy seed in diagnosis of enteric fistulas to various organs. Both methods will be used in the same patient. Diagnostic performance of both methods will be compared in terms of sensitivity, specifity, positive and negative predictive values.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study for comparison of computed tomography and oral poppy seed ingestion in fistula (Experimental): Single arm study for comparison of computed tomography and oral poppy seed ingestion in fistula diagnosis.
  Interventions: Diagnostic Test: computed tomography and poppy seed

INTERVENTIONS:
Diagnostic Test: computed tomography and poppy seed — comparison of both interventions
  Other Names: computed tomography; oral poppy seed

SUMMARY:
Primary objective of the present study is to compare the diagnostic efficacy of oral poppy seed ingestion versus the classic abdominopelvic computed tomography scan with oral, ıntravenous and rectal contrast in diagnosis of gastrointestinal fistulas in gynecologic oncology practice.

DETAILED DESCRIPTION:
Gastrointestinal fistulas are pathologic epithelial bridgings and connections between various loops or intestines and abdominal cavity, bladder, vagina, skin or any other organ. Fistulas are potentially dangerous since they may cause electrolyte imbalance, sepsis and abscesses and malnutrition. However, their diagnosis may not be easy since the sensitivity of the abdominopelvic computed tomography scan with oral, ıntravenous and rectal contrast is around 60% percent which is low for such an life threatening emergency. In gynecologic oncology large and small intestine procedures including resection and anastomoses are frequently performed. These procedures may rise suspicions the integrity of anastomoses and may lead to dilemma to intervene or not in case of a diversion from usual clinical progress. Poppy seed ( pappaver somniferum) is a small (about 1 mm each), non digestible cultivable plant seed used in various foods. It is innocent and does not contain any opium or related ingredient. When ingested with yogurt or soup in small amounts it is not absorbed or ingested within intestine and appears as small gray-blue small spheric seed in abdominal drains, vaginal fluid, urine or skin depending on the fistula formation. Poppy seed was first used in diagnosis of intestinal fistulas by Lippert et al. in 1984. Various studies followed in various fields of surgical medicine. However, there have been no reported studies using poppy seen in diagnosis of enteric fistulas in gynecologic oncology practice.

The aim of the present study is to compare the diagnostic efficacy of orally ingested poppy seed and computed tomography in diagnosis of fistulas related to gynecologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* pre and postsurgical gynecologic oncology patients who were suspected to have fistulas connecting gastrointestinal system and skin, bladder, vagina.

Exclusion Criteria:

None

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — gynecologic oncology patients
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
sensitivity, specificity | Two years
  A single arm study that will compare computed tomography and oral poppy seed in diagnosis of enteric fistulas to various organs. Both methods will be used in the same patient.
positive and negative predictive values | Two years
  A single arm study that will compare computed tomography and oral poppy seed in diagnosis of enteric fistulas to various organs. Both methods will be used in the same patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Med Fac Dept. of Obstet and Gynecol. Division of Gynecologic Oncology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zizzo M, Tumiati D, Bassi MC, Zanelli M, Sanguedolce F, Porpiglia F, Fiori C, Campobasso D, Castro Ruiz C, Bergamaschi FA, Maestroni UV, Carrieri G, Cormio L, Biolchini F, Palicelli A, Soriano A, Sassatelli R, Ascani S, Annessi V, Giunta A. Management of colovesical fistula: a systematic review. Minerva Urol Nephrol. 2022 Aug;74(4):400-408. doi: 10.23736/S2724-6051.21.04750-9. Epub 2021 Nov 18. PMID 34791866
- [Result] Schwaibold H, Popiel C, Geist E, Hartung R. Oral intake of poppy seed: a reliable and simple method for diagnosing vesico-enteric fistula. J Urol. 2001 Aug;166(2):530-1. doi: 10.1016/s0022-5347(05)65976-9. PMID 11458060
- [Result] Melchior S, Cudovic D, Jones J, Thomas C, Gillitzer R, Thuroff J. Diagnosis and surgical management of colovesical fistulas due to sigmoid diverticulitis. J Urol. 2009 Sep;182(3):978-82. doi: 10.1016/j.juro.2009.05.022. Epub 2009 Jul 18. PMID 19616793
- [Result] Wensky H, Jongen J. Diagnosis of enterovesical fistula using poppy seeds. Colorectal Dis. 2006 Jan;8(1):71-2. doi: 10.1111/j.1463-1318.2005.00902.x. No abstract available. PMID 16519642
- [Result] Kwon EO, Armenakas NA, Scharf SC, Panagopoulos G, Fracchia JA. The poppy seed test for colovesical fistula: big bang, little bucks! J Urol. 2008 Apr;179(4):1425-7. doi: 10.1016/j.juro.2007.11.085. Epub 2008 Mar 4. PMID 18289575